CLINICAL TRIAL: NCT07215819
Title: Cervical Sagittal Alignment and Its Association With Disability and Neck Awareness in Patients With Chronic Neck Pain
Brief Title: Cervical Sagittal Alignment and Clinical Outcomes in Chronic Neck Pain
Status: Recruiting | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Dilara Ekici Zincirci, Medical Doctor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: Neck Pain
Record Dates: First submitted 2025-10-02; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Neck Pain; Body Awareness; Neck Disability
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neck Pain Group

SUMMARY:
This observational, cross-sectional study investigates the relationship between cervical sagittal alignment parameters, pain-related disability, and body awareness in patients with chronic neck pain. Adult patients aged 18-50 years who present with neck pain lasting at least 3 months and who have undergone a lateral cervical X-ray within the past 3 months will be included. Cervical sagittal parameters will be measured on radiographs, and participants will complete the Neck Disability Index (NDI) and the Fremantle Neck Awareness Questionnaire to evaluate disability and altered body perception.

DETAILED DESCRIPTION:
Chronic neck pain is a common musculoskeletal problem associated with significant disability and reduced quality of life. Although structural and radiological parameters such as cervical sagittal alignment have been proposed as potential contributors to symptom severity, their association with clinical outcomes remains controversial. Altered body awareness, as assessed by the Fremantle Neck Awareness Questionnaire, represents an additional dimension that may influence symptom persistence and disability in these patients.

The aim of this study is to analyze the relationship between cervical sagittal alignment parameters, pain intensity, disability, and body awareness in patients with chronic neck pain. Eligible participants are adults aged 18-50 years with persistent neck pain for at least three months and who have undergone a lateral cervical X-ray within the last three months. Exclusion criteria include a history of cervical trauma or surgery, neurological or psychiatric disorders, inflammatory or systemic diseases, and conditions such as fibromyalgia or malignancy.

Pain intensity will be assessed using the Visual Analog Scale (VAS), disability with the Neck Disability Index (NDI), and body perception with the Fremantle Neck Awareness Questionnaire. Cervical sagittal alignment parameters will be measured retrospectively from the hospital's PACS system. By correlating radiographic findings with patient-reported outcomes, this study seeks to clarify the clinical relevance of cervical sagittal alignment and provide insight into its potential role in the management of chronic neck pain

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-600 years (inclusive), women and men

Chronic neck pain ≥3 months in duration

Lateral cervical X-ray performed within the past 3 months

Exclusion Criteria:

* History of cervical spine trauma or surgery

Cervical radiculopathy (history or current radicular neck/arm pain)

Systemic conditions: diabetes mellitus, inflammatory rheumatic disease, familial hyperlipidemia, malignancy, or fibromyalgia

Known neurological or psychiatric disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults aged 18-60 years with chronic neck pain of at least 3 months' duration will be recruited. Eligible participants must have undergone lateral cervical X-ray imaging within the past 3 months. Both male and female participants will be included.
  Exclusion criteria are: prior history of cervical trauma or surgery; cervical radiculopathy or previous cervical spine operations; systemic conditions such as diabetes mellitus, inflammatory rheumatic disease, familial hyperlipidemia, malignancy, or fibromyalgia; and presence of known neurological or psychiatric disorders.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | At baseline
Fremantle Neck Awareness Questionnaire (FreNAQ-Neck) | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşçıoğlu Şehir Hastanesi, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Only aggregated and anonymized results will be disseminated through scientific publications.